CLINICAL TRIAL: NCT00519311
Title: RCT of an Intervention to Improve the Health of Adolescents With Intellectual Disability
Brief Title: Health Intervention for Adolescents With Intellectual Disability
Acronym: Ask
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Queensland (Other)
Collaborators: National Health and Medical Research Council, Australia (Other)
Responsible Party: Principal Investigator, Nicholas Lennox, Chief Investigator, The University of Queensland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 401647
Record Dates: First submitted 2007-08-21; First posted 2007-08-22 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2015-05

CONDITIONS: Vision Impairment; Hearing Impairment; Obesity
Keywords: Intellectual disability; Health promotion; RCT
MeSH Terms: conditions — Vision Disorders; Hearing Loss; Obesity; Intellectual Disability

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- School based health intervention (Experimental): Educational intervention based on health diary + health check
  Interventions: Behavioral: Health Intervention Package
- Usual care (No Intervention): Normal school curriculum and usual medical care

INTERVENTIONS:
Behavioral: Health Intervention Package — CHAP and Ask Diary
  Arms: School based health intervention

SUMMARY:
People with intellectual disability die five to twenty years earlier than the general population. They also experience high levels of unrecognised disease and receive inadequate levels of health promotion or screening. Although they comprise 2.7% of our population (502 000 Australians) they receive scant, if any, attention in the health literature.

The barriers to good health for this population include: communication difficulties, impaired recall of significant health information, and inadequate training of health service providers. This project attempts to minimise some of these barriers through the use of a Health Intervention Package. Use of this package has been evaluated in adults, but not in adolescents, with intellectual disability.

The Health Intervention Package includes a comprehensive health review, called the Comprehensive Health Assessment Program (CHAP), which is performed by the adolescent's general practitioner, and a diary, the Ask diary, used to collect and store health information and to enhance health advocacy skills. We specifically aim to test if adolescents with intellectual disability using this package will receive better health screening and prevention (our primary outcomes). We also aim to test if using the package results in improved health advocacy by adolescents with intellectual disability and their parents (our secondary outcomes). The tool should also be acceptable to those involved (another secondary outcome). To investigate these aims we propose a clustered randomised controlled trial, a methodology we have used successfully in two previous trials. We will recruit 1000 adolescents (and their carers and teachers) in Special Education Schools and Special Education Units in Queensland.

The CHAP health review aims to produce shorter-term benefits of improved health screening/promotion and disease detection, such as increased sensory testing, identification of vision or hearing impairment, and improved immunisation rates. The Ask diary is intended to produce longer-term benefits such as improved communication about health matters, improved health advocacy skills, improved health record keeping, and increased health maintenance.

DETAILED DESCRIPTION:
The intervention group of school adolescents will receive the Health Intervention Package (consisting of an Ask diary and a CHAP health review). During the first two terms of school the adolescents will receive their own Ask diary and will be trained in the use of the diary by their teacher. At the end of term two the carers and adolescents will be asked to complete part one of the CHAP tool, which comprises a health history, and make an appointed with their GP to complete a health assessment. After this assessment both the adolescent and the parent will use the Ask diary for all ongoing healthcare matters. The control group will receive their customary educational and medical care.

ELIGIBILITY:
Inclusion Criteria:

* Intellectual disability
* Aged >= 10 years
* Attend Special School or Units of Special Education in Southern Queensland

Exclusion Criteria:

* No intellectual disability
* Not aged >= 10 years
* Do not attend Special School or Unit of Special Education in Southern Queensland

Ages: 10 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 732 (Actual)
Dates: Start 2006-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Level of health promotion | Short term
Disease prevention | Short term
Case finding activities (the identification of new disease) | Short term
Acceptability and usefulness of both the CHAP health review and the ASK Diary | Long term

SECONDARY OUTCOMES:
Appropriate health interventions | Short term
Ongoing maintenance of health care | Long term

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas G Lennox, MBBS, Principal Investigator — The University of Queensland
Locations (1):
- Queensland Centre for Intellectual and Developmental Disability, University of Queensland, Mater Hospital, Brisbane, Queensland, Australia

REFERENCES:
- [Background] Lennox N, Ware R, Carrington S, O'Callaghan M, Williams G, McPherson L, Bain C. Ask: a health advocacy program for adolescents with an intellectual disability: a cluster randomised controlled trial. BMC Public Health. 2012 Sep 7;12:750. doi: 10.1186/1471-2458-12-750. PMID 22958354
- [Result] Doan T, Ware R, McPherson L, van Dooren K, Bain C, Carrington S, Einfeld S, Tonge B, Lennox N. Psychotropic medication use in adolescents with intellectual disability living in the community. Pharmacoepidemiol Drug Saf. 2014 Jan;23(1):69-76. doi: 10.1002/pds.3484. Epub 2013 Aug 8. PMID 23929635
- [Result] Carrington S., Lennox N., O'callaghan M., Mcpherson L. & Selva G. (2014) Promoting self-determination for better health and wellbeing for adolescents who have an intellectual disability. Australasian Journal of Special Education 38 (2), 93-114.
- [Result] Lennox N, McPherson L, Bain C, O'Callaghan M, Carrington S, Ware RS. A health advocacy intervention for adolescents with intellectual disability: a cluster randomized controlled trial. Dev Med Child Neurol. 2016 Dec;58(12):1265-1272. doi: 10.1111/dmcn.13174. Epub 2016 Jun 25. PMID 27343021
- [Result] McPherson L, Ware RS, Carrington S, Lennox N. Enhancing Self-Determination in Health: Results of an RCT of the Ask Project, a School-Based Intervention for Adolescents with Intellectual Disability. J Appl Res Intellect Disabil. 2017 Mar;30(2):360-370. doi: 10.1111/jar.12247. Epub 2016 Feb 12. PMID 26868513
- [Result] Krause S, Ware R, McPherson L, Lennox N, O'Callaghan M. Obesity in adolescents with intellectual disability: Prevalence and associated characteristics. Obes Res Clin Pract. 2016 Sep-Oct;10(5):520-530. doi: 10.1016/j.orcp.2015.10.006. Epub 2015 Nov 11. PMID 26559898
- [Result] Patton KA, Ware R, McPherson L, Emerson E, Lennox N. Parent-Related Stress of Male and Female Carers of Adolescents with Intellectual Disabilities and Carers of Children within the General Population: A Cross-Sectional Comparison. J Appl Res Intellect Disabil. 2018 Jan;31(1):51-61. doi: 10.1111/jar.12292. Epub 2016 Oct 4. PMID 27704663